CLINICAL TRIAL: NCT04925817
Title: 3D Ultrasound Microvessel Imaging for Breast Masses
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 21-002713; NCI-2021-04853 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); P30CA015083 (NIH); R03CA241020 (NIH); 21-002713 (Other: Mayo Clinic Institutional Review Board)
Record Dates: First submitted 2021-05-25; First posted 2021-06-14 (Actual); Last update posted 2024-06-07 (Actual); Status verified 2024-06

CONDITIONS: Breast Carcinoma
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Diagnostic (ultrasound microvessel imaging) (Experimental): Patients undergo 3 D ultrasound microvessel imaging over 45 minutes. Patients' medical records are reviewed.
  Interventions: Other: Electronic Health Record Review; Procedure: Ultrasound Microvessel Imaging

INTERVENTIONS:
Other: Electronic Health Record Review — Medical record reviewed
Procedure: Ultrasound Microvessel Imaging — Undergo 3D ultrasound microvessel imaging
  Other Names: 3D Ultrasound Microvessel Imaging; UMI

SUMMARY:
This early phase I trial studies how well 3D ultrasound microvessel imaging works for the diagnosis of breast mass. The 3D ultrasound microvessel imaging technology demonstrates significantly increased vessel detection sensitivity over conventional doppler methods without the need of using contrast agents. This study may improve cancer diagnosis and reduce unnecessary biopsy on benign tumors.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Optimization of imaging protocol for this new ultrasound technology. II. Investigate the diagnostic performance of the new ultrasound technology using clinically indicated biopsy as the reference standard.

OUTLINE:

Patients undergo 3 dimensional (D) ultrasound microvessel imaging over 45 minutes. Patients' medical records are reviewed.

ELIGIBILITY:
Inclusion Criteria:

* Women with solid breast lesion who are scheduled for a clinically indicated ultrasound-guided biopsy.
* Lesion size of 3 mm or larger.
* Age 18 or greater.

Exclusion Criteria:

* Women with previous breast surgery or breast implant.
* Lacking the capacity to consent.
* Women who are pregnant or lactating.
* Women who are receiving cancer therapy such as chemotherapy or radiation therapy.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2021-08-19 (Actual); Primary Completion 2023-05-18 (Actual); Study Completion 2023-05-18 (Actual)

PRIMARY OUTCOMES:
Ultrasound diagnostic accuracy using McNemar's test | Up to 1 year
  Will be compared between conventional ultrasound (US) and conventional US + 3 dimensional (D) ultrasound microvessel imaging (UMI) using McNemar's test.
Ultrasound parameters sensitivity using McNemar's test | Up to 1 year
  Will include diagnostic performance parameters (sensitivity) calculated based on the BI-RADS score.
Ultrasound parameters specificity using McNemar's test | Up to 1 year
  Diagnostic sensitivity comparison between conventional US versus US + 3D-UMIl using the McNemar's test. Scale = Max 100%, Min 0% - The higher, the better.
Ultrasound parameters positive predictive value using McNemar's test | Up to 1 year
  Will include diagnostic performance parameters (positive predictive value) calculated based on the BI-RADS score. Scale = Max 100%, Min 0% - The higher, the better.
Ultrasound parameters negative predictive value using McNemar's test | Up to 1 year
  Will include diagnostic performance parameters (negative predictive value) calculated based on the BI-RADS score. Scale = Max 100%, Min 0% - The higher, the better. .
Ultrasound parameters accuracy using McNemar's test | Up to 1 year
  Will include diagnostic performance parameters (accuracy) calculated based on the BI-RADS score. Scale = Max 100%, Min 0% - The higher, the better.
Ultrasound parameters calculated by McNemar's test | Up to 1 year
  Will include Data System (BI-RADS) score calculated based on the BI-RADS score. Scale = Max 100%, Min 0% - The higher, the better.
Ultrasound parameters vs. Breast Image Reporting using McNemar's test | Up to 1 year
  Will include Breast Imaging Reporting calculated based on the BI-RADS score. Scale = Max 100%, Min 0% - The higher, the better.

CONTACTS AND LOCATIONS:
Overall Officials: Shigao Chen, Ph.D., Principal Investigator — Mayo Clinic in Rochester
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials

DOCUMENTS (1):
  • Informed Consent Form (2023-03-24): https://cdn.clinicaltrials.gov/large-docs/17/NCT04925817/ICF_000.pdf